CLINICAL TRIAL: NCT01424215
Title: The Use of Fluorescent Imaging for Intraoperative Cholangiogram During Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Danny A Sherwinter, Attending, Surgery, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/08/VA01
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Cholelithiasis; Cholecystitis; Pancreatitis Biliary; Colic of Gallbladder Without Mention of Cholecystitis
MeSH Terms: conditions — Cholelithiasis; Cholecystitis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICG injection with Spyscope imaging (Experimental): Indocyanine Green (ICG)
  Interventions: Drug: Indocyanine Green (ICG)
- Standard Critical View Technique (No Intervention): 50 patients will be randomized to the no treatment arm. These patients will not get ICG injection but rather will have the standard technique for laparoscopic cholecystectomy performed including the critical view technique to expose the important structures prior to clipping and division.

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — Injection of ICG intravenously then intraoperative imaging of the biliary anatomy during laparoscopic cholecystectomy using a near infrared (NIRF) imaging camera(Spy scope, Novadaq Canada)
  Other Names: Spy scope
  Arms: ICG injection with Spyscope imaging

SUMMARY:
The purpose of this study is to evaluate whether a fluorescent die and a special infrared camera can assist with the identification of the important structures during laparoscopic cholecystectomy. This finding may assist surgeons to perform laparoscopic cholecystectomy in less time and in a safer fashion than standard laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether systemically injected ICG, when fluorescing in response to NIR illumination, can assist with the identification of the CBD (common bile duct)during laparoscopic cholecystectomy. This finding may assist surgeons to perform laparoscopic cholecystectomy in less time and with less morbidity than standard laparoscopic cholecystectomy.It is expected that a successful outcome to such a trial will result in less time in the operating room and less morbidity following laparoscopic cholecystectomy.

Laparoscopic cholecystectomy is indicated for cholecystitis, biliary colic, resolved biliary pancreatitis, and symptomatic cholelithiasis. Laparoscopic cholecystectomy involves the introduction of surgical instruments through a number (usually 4) of small incisions measuring about 5-12 mm each with visual guidance being provided by means of a camera attached to an endoscope introduced through a similarly small access port. Laparoscopic techniques offer numerous benefits including a decrease in postoperative pain, some improvement in time to tolerance of food and return of bowel function, shorter hospital stay and more rapid return to normal activity.

Laparoscopic cholecystectomy is one of the most frequently performed surgical procedures in the United States. Iatrogenic bile duct injuries are a serious complication and patients undergoing the laparoscopic type of cholecystectomy are at increased risk for this complication. To minimize risk of injury, techniques such as "critical view" (dissection and visualization of the cystic duct and cystic artery) have been developed. However, adhesions, inflammation and anatomical variation can make surgical dissection and identification of significant structures difficult. In addition significantly longer operative times are seen when attempting to obtain the critical view. Some advocate the routine use of cholangiography (IOC) but the national standard of care remains to only perform IOC selectively. IOC requires cannulation of the cystic duct, injection of iodinated dye, and fluoroscopy which adds significantly to the operative time and morbidity especially in centers where routine IOC is not performed.

The present study will investigate whether the use of NIRF after injection of ICG will make identification of the Biliary structures and CBD clearer and decrease the time required to dissect out critical structures and perform safe cholecystectomy.

The SPY® Intraoperative Imaging System is cleared for use in Canada, Japan, Europe and the US. SPY was originally developed for applications in cardiac surgery and allows cardiac surgeons to visually assess bypass graft quality in real-time while the patient is still in the operating room. Subsequently, SPY has received clearance from the FDA for use in plastic and reconstructive surgery and in solid organ transplant.

The SPY Intraoperative Imaging System was originally developed for open surgical procedures using ICG, which is an FDA approved drug. ICG is a fluorescent compound, which can be administered intravenously or intra-arterially. The dye absorbs light in the near infrared (NIR) region at 806 nm, and emits light at a slightly longer wavelength, 830 nm. When injected intravenously, ICG rapidly and extensively binds to plasma proteins and is confined to the intravascular compartment with minimal leakage into the interstitium under normal conditions. ICG is taken up by the liver and then excreted into the biliary system where it can be imaged. The SPY System has been the subject of numerous peer reviewed publications demonstrating its safety .

SPY scope, the endoscopic version of SPY, is an endoscopic visible (VIS) NIR imaging system consisting of:

1. An endoscopic light source that provides illumination for visible light imaging and NIR fluorescence excitation to the endoscope via a flexible light guide
2. Rigid endoscopes optimized for illuminating the field of view and transmitting images in the visible and NIR spectrum, and
3. A high definition (HD) endoscopic camera system connected to the endoscope eyepiece and acquiring high resolution visible and NIR fluorescence images The ICG (25 mg per vial) will be reconstituted according to the manufacturer's instructions using the entire contents (10 ml) of the sterile diluent supplied, yielding a 2.5 mg/ml solution of ICG or using half of the diluent supplied (5 ml) yielding a 5 mg/ml solution.

ICG Diagnostic Procedure: 3ml of 2.5 mg/ml solution (Akorn product, US Monograph) The ICG may be administered through a peripheral venous access. Based on our prior experience in colorectal cases 1.0 ml of a 2.5 mg/ml solution of ICG (flushed with 10 ml saline) will be administered.

Our study will include patients undergoing laparoscopic cholecystectomy for both acute cholecystitis and non-acute symptomatic cholelithiasis. The standard operating technique will be used for all patients including the critical view technique and fluoroscopic IOC if clinically indicated.

Our primary endpoint will be operative time measured as the time from the beginning of the dissection until the gallbladder is separated entirely from the gall bladder fossa.

Secondary endpoints will be time to identification of structures and safety of the operation. Other endpoints such as CBD injury and postop bile leak will be included if identified.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide an informed consent
* Subject is willing and able to comply with the study procedures
* Subject speaks English and is able to understand the study procedures
* A pregnancy test for women of childbearing potential prior to surgery
* Subject is scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Subject has uremia, serum creatinine >2.5 mg/dl
* Subject has a previous history of adverse reaction or allergy to ICG, iodine, shellfish or iodine dyes
* Subjects in whom the use of x-ray dye or ICG is contraindicated including development of adverse events when previously or presently administered
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Subject is a pregnant or lactating female
* Subject is actively participating in another drug, biologic and/or device protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Derived] Sherwinter DA. Identification of anomolous biliary anatomy using near-infrared cholangiography. J Gastrointest Surg. 2012 Sep;16(9):1814-5. doi: 10.1007/s11605-012-1945-z. Epub 2012 Jul 3. PMID 22752550

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICG Injection With Spyscope Imaging | Standard Critical View Technique
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICG Injection With Spyscope Imaging | Standard Critical View Technique | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 46 | 80
  Male | 16 | 4 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: The primary endpoint will be operative time measured as the minutes from the beginning of the dissection until the gallbladder is separated entirely from the gall bladder fossa. Minutes from start of procedure until recognition of structures.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 48hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ICG Injection With Spyscope Imaging | Standard Critical View Technique
Number analyzed (Participants) | 50 | 50
minutes | 51.6 (11.06) | 44.4 (8.48)

2. Secondary Outcome: Identification of Structures
Description: Minutes Surgeon is able to identify structures.
Time Frame: 0- 14 days Postoeprative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ICG Injection With Spyscope Imaging | Standard Critical View Technique
Number analyzed (Participants) | 50 | 50
minutes | 17.1 (6.05) | 20.2 (7.52)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Mortality
Arm/Group | ICG Injection With Spyscope Imaging | Standard Critical View Technique
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT01424215/Prot_SAP_000.pdf